CLINICAL TRIAL: NCT01841060
Title: Assessment of the Effectiveness of Local Ablathermy Radio Frequency (RF) Bronchial Tumors Primitive Stage IA Non-surgical Patients. Phase II Multicenter National
Brief Title: Assessment of the Effectiveness of Local Ablathermy Radio Frequency Bronchial Tumors Primitive
Acronym: PARF2008
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB2008-34
Record Dates: First submitted 2012-10-29; First posted 2013-04-26 (Estimated); Results first posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Malignant Non-small Cell Neoplasm of Lung Stage Ia
Keywords: Malignant Non-small Cell Neoplasm of Lung
MeSH Terms: interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiofrequency ablathermy (Experimental): Percutaneous radiofrequency ablation (RFA)
  Interventions: Procedure: Percutaneous radiofrequency ablation (RFA)

INTERVENTIONS:
Procedure: Percutaneous radiofrequency ablation (RFA) — Computed tomography (CT) was used to treat tumors under general anesthesia. Thoracic epidural anesthesia was administered in case of contraindication to general anesthesia mostly due to poor respiratory function. All patients were treated with the same multitine electrodes (LeVeen; Boston Scientific, Nattick. MA) measuring 3, 3.5, or 4 cm in diameter and at least 10 mm larger than the diameter of the target tumor. Multiple overlapping ablations were performed, when needed, in different parts of the tumor in order to cover the entire volume.

SUMMARY:
Lung tumors of non-small cell stage 1A are usually treated surgically but many patients are not operable because of their condition or respiratory problems associated with it. The treatment is then suggested that local radiotherapy is conventionally carried out in split mode for 6 weeks at a dose of 60-65 Gy irradiation mode This exposes the patient to complications, including post-radiation pneumonitis.

DETAILED DESCRIPTION:
Lung tumors of non-small cell stage 1A are usually treated surgically but many patients are not operable because of their condition or respiratory problems associated with it.

The treatment is then suggested that local radiotherapy is conventionally carried out in split mode for 6 weeks at a dose of 60-65 Gy irradiation mode This exposes the patient to complications, including post-radiation pneumonitis.

This can be problematic in patients with respiratory failure for which surgical treatment has been challenged. Radiofrequency pulmonary developed as a therapeutic alternative, it has the advantage of being performed in a session with less toxicity in the lung parenchyma

ELIGIBILITY:
Inclusion criteria :

1. Patients over 18 years
2. Histological diagnosis of non-small cell lung tumor established.
3. Stage 1A tumors (lesions <= 3 cm, N0) report prepared by PET and CT
4. Surgical treatment of the lesion contrindiqué or refused by the patient,
5. ARF considered technically feasible after discussing the case in a multidisciplinary meeting (RCP)
6. Expectancy greater than 6 months life
7. PET before inclusion (8 weeks maximum before radiofrequency) showing uptake (SUV> = 2.5) at the lesion to be treated,
8. Signed informed consent,
9. Patient affiliated to a social security scheme.

Exclusion criteria :

1. Location of the lesion does not allow achieving ablathermy under satisfactory conditions: lesion contiguous to the major anatomical structures of the mediastinum, hilar location (less than 1 cm from the hilum)
2. Disorder of uncontrolled bleeding (TP <50% TCA> 1.5 x control).
3. Abnormal blood count platelets <90000/mm3
4. Cons-indication to general anesthesia
5. Patient with a cardiac pacemaker if a review indicates treatment against ARF
6. pregnancy
7. Patient included in another clinical study
8. Unable to undergo medical monitoring test for geographical, social or psychological reasons,
9. Private patient freedom and major subject of a measure of legal protection or unable to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-11; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean PALUSSIERE, MD, Study Chair — Institut Bergonié
Locations (9):
- France (9):
  - CHU de Bordeaux, Bordeaux
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital de Tenon, Paris
  - CH de Pau, Pau
  - CHU de Rennes, Rennes
  - CHU de Strasbourg, Strasbourg
  - CHU Rangueil-Larrey, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Palussiere J, Chomy F, Savina M, Deschamps F, Gaubert JY, Renault A, Bonnefoy O, Laurent F, Meunier C, Bellera C, Mathoulin-Pelissier S, de Baere T. Radiofrequency ablation of stage IA non-small cell lung cancer in patients ineligible for surgery: results of a prospective multicenter phase II trial. J Cardiothorac Surg. 2018 Aug 24;13(1):91. doi: 10.1186/s13019-018-0773-y. PMID 30143031

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Treated With Radiofrequency Ablation (RFA): RFA treatment: Computed tomography (CT) was used to treat tumors under general anesthesia. Thoracic epidural anesthesia was administered in case of contraindication to general anesthesia mostly due to poor respiratory function. All patients were treated with the same multitine electrodes (LeVeen; Boston Scientific, Nattick. MA) measuring 3, 3.5, or 4 cm in diameter and at least 10 mm larger than the diameter of the target tumor. Multiple overlapping ablations were performed, when needed, in different parts of the tumor in order to cover the entire volume.
Period: Overall Study
Arm/Group | Patients Treated With Radiofrequency Ablation (RFA)
Started | 42
Completed | 32
Not Completed | 10
Not completed — Protocol Violation | 10

BASELINE CHARACTERISTICS:
Population: Patients treated with Radiofrequency ablation (RFA)
Arm/Group | Patients Treated With Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 42

OUTCOME MEASURES:

1. Primary Outcome: Local Tumor Control Rate 1 Year After Percutaneous Radiofrequency Ablation (RFA)
Description: local control is defined as the absence of progression of the ablated site. rate is defined as the number of alive patient without local progression divided by the number of patients alive at one year.
Time Frame: one year after percutaneous radiofrequency ablation (RFA)
Population: Patients alive at one year
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Treated With Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 32
Participants | 5

2. Secondary Outcome: Local Tumor Control Rate 3 Years After Percutaneous Radiofrequency Ablation (RFA)
Description: local control is defined as the absence of progression of the ablated site. rate is defined as the number of alive patient without local progression divided by the number of patients alive at thee years.
Time Frame: three years after percutaneous radiofrequency ablation (RFA)
Population: Patients alive at three years
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Treated With Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 16
Participants | 3

3. Secondary Outcome: 1-year Overall Survival (OS) Rate
Description: OS was defined as the time from RFA treatment to death, whatever the cause. If the patient was still alive at the end of study or lost to follow-up, the patient was censored at the date of last news. 1-year overall survival rate was estimated using the Kaplan-Meier estimator.
Time Frame: 1 year after RFA
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Treated With Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 36
Participants | 33

4. Secondary Outcome: 3-year Overall Survival (OS) Rate
Description: OS was defined as the time from RFA treatment to death, whatever the cause. If the patient was still alive at the end of study or lost to follow-up, the patient was censored at the date of last news.
Time Frame: 3 years after RFA
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Treated With Radiofrequency Ablation (RFA)
Number analyzed (Participants) | 36
Participants | 21

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Radiofrequency Ablathermy
All-Cause Mortality (participants affected / at risk) | 15/42
Serious Adverse Events (participants affected / at risk) | 2/42
Other Adverse Events (participants affected / at risk) | 3/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency Ablathermy (N=42)
Thromboembolic event (Vascular disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency Ablathermy (N=42)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
fracture (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes